CLINICAL TRIAL: NCT01460212
Title: Magnetic Resonance Imaging Study of Cognitive-Behavior Therapy for Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chun Wang, The attending physician, Dr., Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QYK09184
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Major Depressive Disorder
Keywords: Cognitive-Behavior Therapy; Magnetic Resonance Imaging; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine; Sertraline; Paroxetine; Citalopram; Escitalopram; Fluvoxamine; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavior Therapy group (Experimental): treatment with Cognitive-Behavior Therapy
  Interventions: Behavioral: Cognitive-Behavior Therapy
- SSRI antidepressants (Active Comparator): treatment by SSRI antidepressant
  Interventions: Drug: SSRI antidepressants

INTERVENTIONS:
Drug: SSRI antidepressants — SSRI antidepressants are Selective serotonin reuptake inhibitors. They include fluoxetine (Prozac); sertraline (Zoloft); paroxetine (Paxil); citalopram (Celexa) ;escitalopram (Lexapro) and fluvoxamine (Luvox). It will be chosen according to special condition of every patient.
  Other Names: fluoxetine (Prozac); sertraline (Zoloft); paroxetine (Paxil); citalopram (Celexa); escitalopram (Lexapro); fluvoxamine (Luvox)
  Arms: SSRI antidepressants
Behavioral: Cognitive-Behavior Therapy — The essence of CBT is a learning process through which an appropriate pattern in cognitive and behavioral could be learn and stored as memory
  Other Names: cognitive behavioural therapy（CBT）
  Arms: Cognitive-Behavior Therapy group

SUMMARY:
Study hypothesis: psychotherapy and SSRI treatment effect in different brain way: psychotherapy in "up to down" way and SSRI in "down to up" way. The investigators will explore this hypothesis in major depressive disorder outpatients with Magnetic Resonance Imaging analysis in this study. Patients in different groups will be treated by psychotherapy or SSRI treatment. They will all be checked with Magnetic Resonance Imaging pro and after 12 weeks of treatment.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria undergo an examination that included a diagnostic interview, vision test, and psychophysiological measures. Participants then undergo the baseline fMRI scan within 48 hours, after that, they will receive psychotherapy or SSRI treatment.and returned the scan once they completed the therapy.

ELIGIBILITY:
Inclusion Criteria:

* meet SCID -Ⅰ/P major depressive disorder diagnosis;
* Right handedness;
* good visual acuity.

Exclusion Criteria:

* neurological disease ;
* serious physical illness (e.g. heart, lung, liver, kidney or blood system disease);
* with other mental disorder;
* psychotic symptoms
* personality disorders;
* pregnancy;
* suicidal risk;
* treatment by antidepressants or other psychotropic medications within 6 months prior to the start of the trial;
* with contraindication for MRI

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAMD) | an expected average of 6 months
  The 24-item version of the Hamilton Rating Scale for Depression (HAMD; Hamilton, 1960) will be used for measuring severity of depressive symptoms. Minimum and maximum possible values are respectively 0 and 78. Lower scores show more mild depression.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging | an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, doctor, Principal Investigator — Nanjing Medical University
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China